CLINICAL TRIAL: NCT06084754
Title: Effect of Pulsed Electromagnetic Field Stimulation on Localized Pediatric Osteomyelitis : Randomized Control Trail Study
Brief Title: Effect of Pulsed Electromagnetic Field Stimulation on Localized Pediatric Osteomyelitis
Acronym: PEMF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Eltayeb, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004589
Record Dates: First submitted 2023-09-19; First posted 2023-10-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; Pulsed Electromagnetic Field
MeSH Terms: conditions — Osteomyelitis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Study group) (Experimental): pulsed electromagnetic field and medical treatment ( vancomycin IV injection 1gm divided 250mg every 6hours )
  Interventions: Device: pulsed electromagnetic field; Drug: Antibiotics
- Group B(control group) (Active Comparator): medical treatment only (vancomycin IV injection 1gm divided 250mg every 6hours )
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Device: pulsed electromagnetic field — pulsed electromagnetic field will be over the site of osteomyelitis where patient in supine lying position. the treatment parameters will be set as10 HZ frequency , 20 gauss amplitude, duration about 120 minutes.
  Other Names: CRYOMAG PROFESSIONAL.LEVEL,s.r.l
  Arms: Group A (Study group)
Drug: Antibiotics — Vancomycin IV injection 1gm divided 250mg every 6hours

SUMMARY:
This study will be applied to evaluate effect of pulsed electromagnetic field on pediatric localized osteomyelitis.

DETAILED DESCRIPTION:
Twenty (11 girls, 9 boys) patients will participate in this study. Their ages ranged from 5 to 16 years. They will randomly divide into two groups. Group A ( study group) will receive pulsed electromagnetic field in addition to medical treatment three times per week for two months , Group B(control group ) will receive medical treatment only.

ELIGIBILITY:
Inclusion Criteria:

1. All patients suffering from localized osteomyelitis in one or both lower limbs
2. All patients will be assessed by a physician before starting the study procedures.

Exclusion Criteria:

1. Patients with immune disorders .
2. Patients who suffer from any systemic diseases that may interfere with the objectives of the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Changing of osteomyelitis signs | pre treatment and post two months of treatment
  through CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Nessrien A. AbdelRashid, Ass.professor, Study Director — physical therapy, Cairo university
Locations (1):
- Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided